CLINICAL TRIAL: NCT01422343
Title: Correlation of Microparticles With Risk of Early Re-stenosis After Percutaneous Transluminal Angioplasty in Patients With Peripheral Arterial Disease
Brief Title: Microparticles and the Risk of Re-stenosis Following Balloon Angioplasty in Patients With Peripheral Arterial Disease
Status: Withdrawn | Type: Observational
Why Stopped: Shortage of personnel / main study initiator no longer available
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Bern (Other)
Responsible Party: Prof. Iris Baumgartner, Bern University Hospital
Other Study IDs: 068/09
Record Dates: First submitted 2011-03-28; First posted 2011-08-23 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-09

CONDITIONS: Peripheral Vascular Diseases
Keywords: peripheral arterial disease; cell-derived microparticles; immunity, innate; blood coagulation
MeSH Terms: conditions — Peripheral Vascular Diseases; Peripheral Arterial Disease; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1
  Interventions: Procedure: percutaneous transluminal angioplasty femoro-popliteal

INTERVENTIONS:
Procedure: percutaneous transluminal angioplasty femoro-popliteal — percutaneous transluminal angioplasty femoro-popliteal

SUMMARY:
Although microparticles have been well-documented as mediators of inflammation and coagulation in various cardio-vascular disease events, it is currently not known how Percutaneous Transluminal Angioplasty (PTA) for peripheral arterial disease influences microparticle numbers, phenotype and distribution pre- and post interventionally and how they are related to or affect the incidence of early re-stenosis - or if indeed they may be used to predict patients at risk of early re-stenosis.

DETAILED DESCRIPTION:
Background

Background and rationale of the study:

Atherosclerosis is an increasing widespread systemic disease, representing a significant cause of morbidity and mortality for those affected by it. Age-adjusted prevalence of peripheral arterial disease lies at 12%, increasing to 20% in persons above the age of 70. Five percent of patients with intermittent claudication develop critical limb ischemia within five years from early symptoms, and are considered to be at risk of major amputation.

Whilst bypass surgery remains a valid treatment option for patients with peripheral arterial disease and ensures good long-term anatomical patency and clinical durability, this trusted surgical procedure comes at a certain risk of morbidity and mortality. Furthermore, patent vessels of good quality, particularly veins needed for the bypass procedure, are often unavailable and impose limitations to the method. Percutaneous transluminal angioplasty (PTA) has evolved in the past years as a valid treatment modality for patients with stenotic arterial lesions of the lower extremities due to peripheral arterial disease. However, re-stenosis following PTA for peripheral arterial disease is not uncommon and poses a serious therapeutic problem. Despite the increasing prevalence and incidence of peripheral arterial disease in the population, timely diagnosis or use of diagnostic and prognostic markers are still lacking (still lags behind the current diagnostic and treatment strategies for coronary artery disease and acute coronary syndromes). Indeed, currently, only few recognisable risk factors for the development of re-stenosis have been recognized. These include beside clinically advanced peripheral arterial disease and diabetes mellitus, also pro-inflammatory and pro-coagulatory states with high CRP and fibrinogen as well as post-interventionally increased levels of von Willebrand factor and plasminogen inhibitor-1. Furthermore, TGF-beta1 levels are also significantly increased in patients with re-stenosis. The actual missing link between these "common" pro-inflammatory markers and the occurrence of re-stenosis is however not known - the answer may lie in subcellular fragments circulating in the blood.

Indeed, these so-called cell-derived plasma microparticles (MPs) are small phospholipid vesicles up to 1.5 µm in size that are released from platelets, circulating leukocytes and endothelial cells upon activation. Originating from lipid rafts, they contain defined bioactive molecules that are potentially implicated in thrombogenesis and trans-cellular activation. Additionally, pro-inflammatory functions may be mediated by putative ligand-receptor interactions, classical pathway complement activation 11 and by triggering or modifying target cells and their functions. Furthermore, MPs represent a population of phosphatidylserine-exposing sub-cellular fragments, function as "carriers" of circulating tissue factor, and may be invaluable in maintaining normal haemostasis when platelet function is impaired. Microparticles transport pro-inflammatory molecules such as interleukins, interferon gamma and tumour necrosis factor alpha. Increasing evidence suggests that released MPs are more than just inert cell debris or irrelevant platelet dust. Instead, they are potent biological agents found in healthy individuals but also implicated in a variety of diseases, including vascular inflammatory states after cardiopulmonary bypass surgery, acute coronary syndromes, and diseases associated with the metabolic syndrome e.g. diabetes mellitus. Patients with peripheral arterial disease (PAD) due to diabetes mellitus type 2 also present with an increased "baseline" pro-inflammatory and pro-coagulatory state. It appears that in diabetic patients platelet-derived microparticles may participate in the development or progression of atherosclerosis. Moreover, elevated numbers of microparticles, specifically platelet-derived, have been described in patients with peripheral arterial disease.

Although microparticles have been well-documented as mediators of inflammation and coagulation in various cardio-vascular disease events, it is currently not known how PTA for peripheral arterial disease influences microparticle numbers, phenotype and distribution pre- and post interventionally and how they are related to or affect the incidence of early re-stenosis - or if indeed they may be used to predict patients at risk of early re-stenosis.

Objective

Hypothesis and Aims:

Hypothesis: Plasma derived microparticles actively influence the course of disease and are associated with early re-stenosis/re-occlusion after angioplasty in patients (men and women) with peripheral arterial disease by acting as mediators between innate- and cellular immunity as well as the coagulation system.

Aim 1: The first aim of the study is to characterise and quantify microparticles from peripheral blood samples at baseline and one day post-angioplasty Aim 2: The second aim is to characterise and quantify microparticles in the follow up period 2 weeks, 3 and 6 months post-angioplasty and to identify whether the microparticle profile can be used to define patients at greater risk for re-stenosis.

Aim 3: The third aim is to address the possible gender differences in microparticle distribution and numbers in a sub-group analysis. This will be an important part of the project as currently no such data exist.

Methods

Study design: The study will include measurements at baseline, one day, 2 weeks, 3 and 6 months post-angioplasty.

Evaluation Obtain informed consent: day (d)0 Physical examination: d0, d+1, 2 weeks, 3 and 6 months post-intervention Ankle-brachial index (ABI) measurement: d0, d+1, 2 weeks, 3 and 6 months post-intervention Duplex sonography: 6 months post-intervention Angioplasty: d0 (begin of study Blood sampling routine*: d0, d+1 Blood sampling study**: d0, d+1, 2 weeks, 3 and 6 months post-intervention

* Fasting glucose, HBA1c, lipid profile, creatinine, haemoglobin, leukocyte profile, thrombocytes, C-reactive protein

** Microparticles, cytokines, complement (=5ml serum, 2.7ml EDTA plasma, 10ml citrate)

ELIGIBILITY:
Inclusion Criteria:

* male or female
* 60-85 years
* femoro-popliteal stenosis
* TASC B or C category
* HBA1c <9%, if diabetic
* creatinine <130µg/ml
* blood pressure <160/95mmHg
* thrombocyte aggregation inhibitors or coumarine derivatives

Exclusion Criteria

* <60 or >85 years
* stenosis not in femoro-popliteal axis
* TASC A or D category
* HBA1c >9%, if diabetic
* creatinine >130µg/ml
* blood pressure >160/95mmHg
* major trauma
* malignancy
* anti-phospholipid syndrome
* relevant hepatic disease
* major operation within 1 month of enrolment

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients (male and female) with peripheral arterial disease presenting at the angiology clinic, Bern University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-05; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Number of participants with early re-stenosis post-angioplasty | 6 month post-angioplasty

SECONDARY OUTCOMES:
Number of and changes in circulating cell-derived microparticles, measured by flow cytometric analysis of peripheral blood samples, and correlation with early re-stenosis post-PTA | 6 months post-angioplasty

CONTACTS AND LOCATIONS:
Overall Officials: Iris Baumgartner, DMD, Principal Investigator — Bern University Hospital

REFERENCES:
- [Background] Dormandy JA, Rutherford RB. Management of peripheral arterial disease (PAD). TASC Working Group. TransAtlantic Inter-Society Consensus (TASC). J Vasc Surg. 2000 Jan;31(1 Pt 2):S1-S296. No abstract available. PMID 10666287
- [Background] Nieuwland R, Berckmans RJ, Rotteveel-Eijkman RC, Maquelin KN, Roozendaal KJ, Jansen PG, ten Have K, Eijsman L, Hack CE, Sturk A. Cell-derived microparticles generated in patients during cardiopulmonary bypass are highly procoagulant. Circulation. 1997 Nov 18;96(10):3534-41. doi: 10.1161/01.cir.96.10.3534. PMID 9396452
- [Background] Mallat Z, Benamer H, Hugel B, Benessiano J, Steg PG, Freyssinet JM, Tedgui A. Elevated levels of shed membrane microparticles with procoagulant potential in the peripheral circulating blood of patients with acute coronary syndromes. Circulation. 2000 Feb 29;101(8):841-3. doi: 10.1161/01.cir.101.8.841. PMID 10694520
- [Background] Diamant M, Nieuwland R, Pablo RF, Sturk A, Smit JW, Radder JK. Elevated numbers of tissue-factor exposing microparticles correlate with components of the metabolic syndrome in uncomplicated type 2 diabetes mellitus. Circulation. 2002 Nov 5;106(19):2442-7. doi: 10.1161/01.cir.0000036596.59665.c6. PMID 12417540